CLINICAL TRIAL: NCT03219294
Title: Does Deep Neuromuscular Blockade Improve Operating Conditions During Total Hip Replacements?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Craig Curry (Other)
Collaborators: MaineHealth (Other); Spectrum Medical Group Anesthesiology (Other)
Responsible Party: Sponsor-Investigator, Craig Curry, Anesthesiologist, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 988210-2
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Arthropathy of Hip
Keywords: neuromuscular blockade; sugammadex
MeSH Terms: interventions — Vecuronium Bromide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologist will NOT be blinded, but the orthopedic surgeon performing the hip replacement surgery will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Neuromuscular Blockade (NMB) (Active Comparator): Intubating dose of Vecuronium 0.1 mg/kg (IBW) and re-dosing with 0.0125 to 0.05 mg/kg as needed to achieve and maintain 1 to 2 train-of-four (TOF) contractions. Redosing in this manner is a current clinical practice.
  Interventions: Drug: Vecuronium 0.1 mg/kg
- Deep NMB (Active Comparator): Deep NMB: Intubating dose of Vecuronium 0.2 mg/kg (IBW) and re-dosing with 0.025 to 0.1 mg/kg to achieve and maintain zero twitches in the TOF, and post tetanic count (PTC) of 1 to 2 contractions. This level of blockade is new to the practice since approval of the drug for use at Maine Medical Center (MMC) but is in common use since the advent of Sugammadex.
  Interventions: Drug: Vecuronium 0.2mg/kg

INTERVENTIONS:
Drug: Vecuronium 0.1 mg/kg — Vecuronium will be administered to achieve and maintain 1 to 2 TOF contractions.
  Other Names: vecuronium bromide
  Arms: Moderate Neuromuscular Blockade (NMB)
Drug: Vecuronium 0.2mg/kg — Vecuronium will be administered to achieve and 0 TOF/PTC 1-2.
  Other Names: vecuronium bromide
  Arms: Deep NMB

SUMMARY:
During many surgeries, increased muscle tension makes it harder for the surgeon to expose the site of surgery and work within the incision. Neuromuscular blockade (NMB) drugs such as Vecuronium bind to neurotransmitter (acetyl choline) receptors at the neuromuscular junction, blocking their action and producing muscle relaxation. This muscle relaxation allows easier retraction of muscle tissues and manipulation of structures in the wound. Improved surgical conditions are likely to result in improved patient outcomes. While increased depths of NMB have been shown to optimize surgical conditions during intra-abdominal and retroperitoneal procedures, the impact of NMB depth has not been reported for orthopedic surgeries.1 To address this, we propose to study the effect of NMB depth on surgical conditions during total hip replacement (THR).

DETAILED DESCRIPTION:
Specific Aims

1. Assess difference in surgical conditions between moderate and deep NMB groups. Enrolled patients will be randomized to receive moderate (n=58) or deep (n=58) NMB. Difference in surgical conditions will be evaluated by:

   1. The number of requests from the surgeon for additional relaxation (NMB) during the procedure. At any time during the operation if the surgeon feels the muscle tension is interfering with ease of operation he will ask for additional muscle relaxation. If the patient is moderately relaxed they will be converted to deep relaxation with additional muscle relaxants. If they are already deeply relaxed no additional relaxants will be administered (as is our current practice). All requests will be recorded.
   2. Rating by the surgeon after each surgery using an internally developed satisfaction scale. The scale was developed by modifying a scale used in a previous study of muscle relaxation in intra-abdominal surgery1 to specify two key elements identified by our surgeon: ease of muscle retraction and femur manipulation.
2. Assess the impact of deep vs moderate NMB on time of surgery, measured from the time of incision to joint reduction.

SIGNIFICANCE If we identify improved surgical conditions with deeper relaxation we will incorporate deep NMB into our routine anesthesia practice for THR.

Vecuronium will be used as NMB drug in all study patients; this agent is currently used in over 90% of THR cases at Maine Medical Center (MMC). As is currently routine Vecuronium will be given after initiation of general anesthesia with propofol to facilitate intubation and further doses of Vecuronium will be given throughout the case as noted below to maintain NMB at the desired depth until the femoral implant is reduced. After the intubating dose of Vecuronium, NMB depth will be monitored every 5 minutes and dosing will be adjusted as needed to maintain a constant depth of NMB according to our current routine practice.

Group 1: Moderate NMB: Intubating dose of Vecuronium of 0.1 mg/kg (IBW) and re-dosing with 0.0125 to 0.05 mg/kg as needed to achieve and maintain 1 to 2 train of four (TOF) contractions. Redosing in this manner is a current clinical practice.

Group 2: Deep NMB: Intubating dose of Vecuronium of 0.2 mg/kg (IBW) and re-dosing with 0.025 to 0.1 mg/kg to achieve and maintain zero twitches in the TOF, and post tetanic count (PTC) of 1 to 2 contractions. This level of blockade is new to the practice since approval of the drug for use at MMC but is in common use since the advent of Sugammadex.

The surgeon may request additional relaxation at anytime for inadequate surgical conditions thought to be related to muscle tension. All requests will be recorded. Patients in the moderate NMB group will receive additional doses of vecuronium to achieve deep NMB (PTC of 1- 2). In the deep NMB group with PTC of 1-2, a saline dose without NMB will be given.

NMB reversal Sugammadex will be given for reversal of NMB after the prosthesis has been reduced, using routine dosing of 2 mg/kg for the moderate group and 4 mg/kg for the deep group, per package insert by Merck.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical status 1-3
* age 50-75
* English speaking
* able to provide informed consent
* BMI equal to less than 30
* non-emergent THR by anterolateral minimally invasive non-cemented total hip arthroplasty

Exclusion Criteria:

* Revision surgery
* Bilateral THR
* ASA 4+
* age less than 50 or greater than 75
* BMI greater than 30
* unable to provide informed consent
* women taking oral contraceptives (Sugammadex used for reversal interferes with their efficacy
* contraindications to general inhalation anesthesia (such as malignant hyperthermia)
* contraindications to NMB (known allergy to NMB)
* chronic kidney disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Curry, MD, Principal Investigator — Maine Medical Center/Spectrum Medical Group
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basad E, Ishaque B, Sturz H, Jerosch J. The anterolateral minimally invasive approach for total hip arthroplasty: technique, pitfalls, and way out. Orthop Clin North Am. 2009 Oct;40(4):473-8, viii. doi: 10.1016/j.ocl.2009.05.001. PMID 19773052
- [Background] Brueckmann B, Sasaki N, Grobara P, Li MK, Woo T, de Bie J, Maktabi M, Lee J, Kwo J, Pino R, Sabouri AS, McGovern F, Staehr-Rye AK, Eikermann M. Effects of sugammadex on incidence of postoperative residual neuromuscular blockade: a randomized, controlled study. Br J Anaesth. 2015 Nov;115(5):743-51. doi: 10.1093/bja/aev104. Epub 2015 May 2. PMID 25935840
- [Background] Madsen MV, Staehr-Rye AK, Gatke MR, Claudius C. Neuromuscular blockade for optimising surgical conditions during abdominal and gynaecological surgery: a systematic review. Acta Anaesthesiol Scand. 2015 Jan;59(1):1-16. doi: 10.1111/aas.12419. Epub 2014 Oct 19. PMID 25328055
- [Background] Paton F, Paulden M, Chambers D, Heirs M, Duffy S, Hunter JM, Sculpher M, Woolacott N. Sugammadex compared with neostigmine/glycopyrrolate for routine reversal of neuromuscular block: a systematic review and economic evaluation. Br J Anaesth. 2010 Nov;105(5):558-67. doi: 10.1093/bja/aeq269. Epub 2010 Oct 8. PMID 20935005
- [Background] Chambers D, Paulden M, Paton F, Heirs M, Duffy S, Craig D, Hunter J, Wilson J, Sculpher M, Woolacott N. Sugammadex for the reversal of muscle relaxation in general anaesthesia: a systematic review and economic assessment. Health Technol Assess. 2010 Jul;14(39):1-211. doi: 10.3310/hta14390. PMID 20688009

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate NMB: Intubating dose of Vecuronium 0.1 mg/kg (IBW) and re-dosing with 0.0125 to 0.05 mg/kg as needed to achieve and maintain 1 to 2 TOF contractions. Redosing in this manner is a current clinical practice.
  Vecuronium 0.1 mg/kg: Vecuronium will be administered to achieve and maintain 1 to 2 TOF contractions.
- Deep NMB: Deep NMB: Intubating dose of Vecuronium 0.2 mg/kg (IBW) and re-dosing with 0.025 to 0.1 mg/kg to achieve and maintain zero twitches in the TOF, and post tetanic count (PTC) of 1 to 2 contractions. This level of blockade is new to the practice since approval of the drug for use at MMC but is in common use since the advent of Sugammadex.
  Vecuronium 0.2mg/kg: Vecuronium will be administered to achieve and 0 TOF/PTC 1-2.
Period: Overall Study
Arm/Group | Moderate NMB | Deep NMB
Started | 58 | 58
Completed | 58 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate NMB | Deep NMB | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (6.7) | 62.9 (7.4) | 63 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 29 | 28 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: Surgical Conditions
Description: The surgeon graded the overall surgical conditions on a 5 point Likert scale, that was taken into account along with requests for additional muscle relaxation. The Likert scale went from 1 (extremely poor conditions: muscles resistant to retraction and obscure view, implant difficult to insert into socket, requires assist) to 5 (optimal conditions: muscles relaxed, excellent view, implant easy to insert).
Time Frame: Through study completion, an average of 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate NMB | Deep NMB
Number analyzed (Participants) | 58 | 58
Participants
  Extremely Poor Conditions | 1 | 2
  Poor Conditions | 11 | 10
  Acceptable Conditions | 30 | 29
  Good Conditions | 15 | 15
  Optimal Conditions | 1 | 2

2. Secondary Outcome: Duration of Surgery
Description: Time from incision to joint reduction
Time Frame: Through study completion, an average of 24 hours for each patient and up to one year for the whole study.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Moderate NMB | Deep NMB
Number analyzed (Participants) | 58 | 58
minutes | 32.6 (1.2) | 33.8 (1.2)

ADVERSE EVENTS:
Time Frame: Patients were monitored for the duration of their surgical case and time in the post-anesthesia care unit until discharge from the hospital, usually 24 hours, and had a post-surgical follow-up several weeks after discharge.
Arm/Group | Moderate NMB | Deep NMB
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03219294/Prot_SAP_001.pdf